CLINICAL TRIAL: NCT06282523
Title: Healthy Minds Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1773; A171600 (Other: UW- Madison); EDUC/COUNSELING PSYCH (Other: UW- Madison); Protocol Version 12/27/23 (Other: UW- Madison)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Depression; Anxiety; Depression/Anxiety
Keywords: meditation; mindfulness
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Minds Program (HMP) - Awareness first (Experimental): Participants will be assigned to use the HMP mobile app on symptoms of psychological distress, and will complete the Awareness module first.
  Interventions: Behavioral: HMP app
- Healthy Minds Research Platform (HMRP) - Awareness first (Experimental): Participants will be assigned to use the HMRP web app on symptoms of psychological distress, and will complete the Awareness module first.
  Interventions: Behavioral: HMRP web app
- HMP - Connection first (Experimental): Participants will be assigned to use the HMP mobile app on symptoms of psychological distress, and will complete the Connection module first.
  Interventions: Behavioral: HMP app
- HMRP - Connection first (Experimental): Participants will be assigned to use the HMRP web app on symptoms of psychological distress, and will complete the Connection module first.
  Interventions: Behavioral: HMRP web app

INTERVENTIONS:
Behavioral: HMP app — The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose.
  Arms: HMP - Connection first; Healthy Minds Program (HMP) - Awareness first
Behavioral: HMRP web app — The HMRP web app is a meditation-based web-based app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMRP provides core content, with instruction administered through a curriculum of guided practices. HMRP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose.
  Arms: HMRP - Connection first; Healthy Minds Research Platform (HMRP) - Awareness first

SUMMARY:
The goal of this clinical trial is to understand the difference between two versions of the Healthy Minds application, a digital well-being program. The main question it aims to answer is the differences between versions of the Healthy Minds application and their effects on well-being.

Participants will complete an online four-week well-being program and complete surveys sent to their email. Participants can expect to participate in the study for four months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Elevated symptoms of depression and anxiety
* Proficient in English
* Access to a smartphone

Exclusion Criteria:

* Prior experience with meditation generally
* Prior use of the Healthy Minds application
* History of psychosis or mania
* Alcohol and/or substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Composite of Patient-Reported Outcomes Measurement Information System (PROMIS) Depression and PROMIS Anxiety | Baseline, weeks 1, 2, 3, 4, and 3 months
  Psychological distress will be computed as a composite of the PROMIS Depression and PROMIS Anxiety measures. We will use the computer adaptive version of both measures which have a mean of 50 and a standard deviation of 10. A composite will be computed by average across T-scores. T-scores range from 10 to 90 with higher scores indicating higher depression or anxiety.

SECONDARY OUTCOMES:
HMP App Utilization: Days | Study duration (4 weeks)
  Number of days the app was accessed.
HMP App Utilization: Number of Activities | Study duration (4 weeks)
  Number of activities completed
HMP App Utilization: Minutes | Study duration (4 weeks)
  Minutes of meditation practice completed
Change in Healthy Minds Index (HM Index): Awareness | Baseline, weeks 1, 2, 3, 4, and 3 months
  The HM Index assesses qualities trained in the HMP and HMRP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. There are 4 awareness items. Mean item scores are reported with a range from 0 to 4 where higher scores indicate more awareness.
Change in Healthy Minds Index (HM Index): Connection | Baseline, weeks 1, 2, 3, 4, and 3 months
  The HM Index assesses qualities trained in the HMP and HMRP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. There are 6 connection items. Mean item scores are reported with a range from 0 to 4 where higher scores indicate more connection.
Change in Healthy Minds Index (HM Index): Purpose | Baseline, weeks 1, 2, 3, 4, and 3 months
  The HM Index assesses qualities trained in the HMP and HMRP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. There are 4 purpose items. Mean item scores are reported with a range from 0 to 4 where higher scores indicate more purpose.
Change in Healthy Minds Index (HM Index): Insight | Baseline, weeks 1, 2, 3, 4, and 3 months
  The HM Index assesses qualities trained in the HMP and HMRP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. There are 3 insight items. Mean item scores are reported with a range from 0 to 4 where higher scores indicate more insight.
Change in Subjective Happiness Scale | Baseline, weeks 1, 2, 3, 4, and 3 months
  The SHS is a 4-item scale of global subjective happiness. It is scored on a 1- to 7-point Likert scale where 1 = less happy and 7 = more happy. Mean scores are reported for a range from 4 to 28 where higher scores indicate more happiness.
Change in Satisfaction with Life Scale (SWLS) | Baseline, weeks 1, 2, 3, 4, and 3 months
  The SWLS is a 5-item scale of subjective satisfaction with life. It is scored on a 1- to 7-point Likert scale where 1 = strongly disagree and 7 = strongly agree. Mean scores are reported for a range from 5 to 35 where higher scores indicate greater satisfaction.
Change in Perceived Stress Scale (PSS-10) | Baseline, weeks 1, 2, 3, 4, and 3 months
  The PSS-10 is a 10-item scale assessing perceived stress. It is scored on a 0- to 4-point Likert scale where 0 = never and 4 = very often. Mean scores are reported for a range from 0 to 40 where higher scores indicate greater stress.
Change in Flourishing Measure | Baseline, weeks 1, 2, 3, 4, and 3 months
  This is a 12-item questionnaire used to assess various domains of flourishing, or human well-being. It is scored on a 0- to 10-point Likert scale where 0 = poor and 10 = excellent. Mean scores are reported for a range from 0 to 120 where higher scores indicate greater human well-being.
Change in Digital Working Alliance Inventory (DWAI) | Baseline, weeks 1, 2, 3, 4, and 3 months
  The DWAI is a 6-item questionnaire assessing participants' alliance with the HMP and HMRP app. It is scored on a 1- to 7-point Likert scale where 1 = strongly disagree and 7 = strongly agree. Total scores range from 6 to 42 where higher scores indicate a stronger working alliance.
Change in Experiences Questionnaire (EQ) Decentering Subscale | Baseline, weeks 1, 2, 3, 4, and 3 months
  Experiences Questionnaire Decentering is an 11-item questionnaire assessing the psychological capacity of decentering. It is scored on a 1- to 5-point Likert scale where 1 = never and 5 = all the time. Mean scores are reported for a total range from 1 to 5 where higher scores indicate more decentering.
Change in Five Facet Mindfulness Questionnaire (FFMQ) Awareness Subscale | Baseline, weeks 1, 2, 3, 4, and 3 months
  FFMQ Awareness is a 8-item questionnaire assessing mindful awareness. It is scored on a 1- to 5-point Likert scale where 1 = never or very rarely true and 5 = very often or always true. Mean scores are reported with a range from 1 to 5 where higher scores indicate more mindful awareness.
Change in NIH Toolbox Loneliness | Baseline, weeks 1, 2, 3, 4, and 3 months
  NIH Toolbox Loneliness is a 5-item questionnaire assessing loneliness. It is scored on a 1- to 5-point Likert scale where 1 = never and 5 = always. Mean scores are reported for a range from 1 to 5 where higher scores indicate more loneliness.
Change in Wellbeing Growth Mindset | Baseline, weeks 1, 2, 3, 4, and 3 months
  Well-being Growth Mindset is a 3-item questionnaire assessing participants' perception of the malleability of wellbeing. It is scored on a 1- to 6-point Likert scale where 1 = strongly disagree and 6 = strongly agree. Total scores range from 3 to 18 where higher scores indicate more of a growth mindset (i.e., wellbeing is malleable).
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Meaning and Purpose | Baseline, weeks 1, 2, 3, 4, and 3 months
  PROMIS Meaning and Purpose is a 37-item questionnaire assessing sense of meaning and purpose. It is scored on a 1- to 5-point Likert scale where 1 = not at all and 5 = very much. Mean scores are reported for a range from 37 to 185 where higher scores indicate greater sense of meaning and purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT06282523/ICF_000.pdf